CLINICAL TRIAL: NCT06142383
Title: A Multi-center, Randomized, Placebo- and Active-controlled, Parallel-group, 24-week Proof of Concept and Dose-finding Study to Evaluate Efficacy, Safety, and Tolerability of XXB750 in Patients With Heart Failure
Brief Title: A Proof of Concept and Dose-finding Study of XXB750 in Patients With Heart Failure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CXXB750A12201; 2023-504678-39-00 (Other: EU CTIS)
Record Dates: First submitted 2023-11-16; First posted 2023-11-21 (Actual); Results first posted 2025-12-24 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
Keywords: Heart failure; randomized; double-blind; dose finding; XXB750
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Patients received either active XXB750 injection or a placebo injection that looks identical to the active injection. Sacubitril/valsartan was administered in an open-label fashion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm 1 (Placebo Comparator): XXB750 Placebo
  Interventions: Biological: Placebo
- Arm 2 (Experimental): XXB750 60 mg
  Interventions: Biological: XXB750 Low dose
- Arm 3 (Experimental): XXB750 120 mg
  Interventions: Biological: XXB750 Medium Dose
- Arm 4 (Experimental): XXB750 240 mg
  Interventions: Biological: XXB750 High Dose
- Arm 5 (Active Comparator): Sacubitril/valsartan, open label tablet, 97/103 mg bid (Sac/Val)
  Interventions: Drug: Sacubitril/valsartan

INTERVENTIONS:
Biological: Placebo — S.C. Injection
  Arms: Arm 1
Biological: XXB750 Low dose — S.C. Injection
  Arms: Arm 2
Biological: XXB750 Medium Dose — S.C. Injection
  Arms: Arm 3
Biological: XXB750 High Dose — S.C. Injection
  Arms: Arm 4
Drug: Sacubitril/valsartan — Tablet
  Arms: Arm 5

SUMMARY:
This was a multicenter, randomized, placebo- and active-controlled, parallel-group, 24-week trial to investigate the efficacy, safety, and tolerability of XXB750 in participants with HFrEF/HFmrEF.

DETAILED DESCRIPTION:
Eligible participants were randomized to receive either subcutaneous (s.c.) XXB750 or placebo; or sacubitril/valsartan for 16 weeks, and then followed-up for 8 weeks.

The study planned to randomize adult participants with LVEF < 50% receiving ACEI/ARB/ARNI and guideline-recommended HF therapies for HFrEF or HFmrEF to three XXB750 target dose levels; a cohort of participants treated with ACEI/ARB before the study was randomized to be converted to open-label sacubitril/valsartan in place of their pre-study ACEI/ARB. A total of 720 participants were planned to be randomized in this study.

Due to safety concerns, in August 2024 the study was halted and dosing of all double-blind injectable medication of XXB750 and matching Placebo was suspended until further notice. All randomized participants actively involved in the study continued to attend study visits as per the study schedule and underwent all study procedures. This included safety, pharmacokinetic, antidrug antibody, and biomarker biological sample collections, physical examinations, and reporting of adverse events. As directed above, injectable study medication (i.e., XXB750 and its matching Placebo) was not administered. On 26-Sep-2024, Novartis made the decision to terminate the study due to safety findings and DMC recommendation.

Due to the early study termination, all participants who had been randomized to receive XXB750 or Placebo were followed up for 12 weeks after they received the last dose which is in accordance with the originally planned follow-up duration as per protocol. Participants who were randomized to the open-label treatment arm 5 and received sacubitril/valsartan as study medication were not further followed up after discontinuation of the open-label study medication. Sacubitril/valsartan is authorized in all participating countries and was, within this study, used as a comparator within the respective labels only. Hence, an additional follow-up for the safety of the participants was not performed; and the investigator could treat the participant with standard-of-care treatment (which includes sacubitril/valsartan) as per his/her clinical judgment.

To help guard the safety of study participants, randomization initially excluded the planned highest target dose of 240 mg XXB750 (i.e., arm 4). The study was terminated prematurely prior to the pre-planned early safety analysis due to an imbalance in worsening heart failure events among participants randomized to XXB750 60 mg and 120 mg. Thus, no participants were exposed to the planned highest target dose of 240 mg every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Current symptom(s) of HF NYHA class II-III and LVEF < 50%
* Elevated NT-proBNP levels at screening.
* Receiving standard of care background HF therapy.

Exclusion Criteria:

* Current acute decompensated HF or hospitalization for HF within 3 months prior to screening.
* Current symptomatic hypotension (for example dizziness/presyncope).
* K+ > 5.4 mmol/L at screening
* eGFR < 30 mL/min/1.73m2 at screening

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (59):
- United States (14):
  - SEC Clinical Research, Dothan, Alabama
  - Heart Center Research Llc, Huntsville, Alabama
  - Nature Coast Clinical Research LLC, Inverness, Florida
  - Inpatient Research Clinical LLC, Miami Lakes, Florida
  - Cardiology Partners Clinical Research Institute, Wellington, Florida
  - American Clinical Trials, Acworth, Georgia
  - The Research Group, Lexington, Kentucky
  - Heart Clinic of Hammond, Hammond, Louisiana
  - Anderson Medical Research, Ft. Washington, Maryland
  - Revival Research Institute, Troy, Michigan
  - Aultman Hospital, Canton, Ohio
  - NexGen Research, Lima, Ohio
  - Tennessee Center For Clinical Trials, Tullahoma, Tennessee
  - Dominion Medical Associates, Richmond, Virginia
- Bulgaria (7):
  - Novartis Investigative Site, Blagoevgrad
  - Novartis Investigative Site, Gabrovo
  - Novartis Investigative Site, Kyustendil
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
- Novartis Investigative Site, Xian, Shanxi, China
- Germany (7):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Gladbeck
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, Papenburg
  - Novartis Investigative Site, Schwäbisch Hall
- Hungary (2):
  - Novartis Investigative Site, Budapest, Pest County
  - Novartis Investigative Site, Balatonfüred
- India (2):
  - Novartis Investigative Site, Belagavi, Karnataka
  - Novartis Investigative Site, Bikaner, Rajasthan
- Italy (6):
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Messina, ME
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Pordenone, PN
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Trieste, TS
- Japan (4):
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Sagamihara, Kanagawa
  - Novartis Investigative Site, Matsumoto, Nagano
- Portugal (2):
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Vila Nova de Gaia
- Slovakia (6):
  - Novartis Investigative Site, Bardejov, Slovakia
  - Novartis Investigative Site, Košice, Slovakia
  - Novartis Investigative Site, Martin, Slovakia
  - Novartis Investigative Site, Nitra, Slovakia
  - Novartis Investigative Site, Prešov, Slovakia
  - Novartis Investigative Site, Svidník, Slovakia
- Spain (7):
  - Novartis Investigative Site, Santiago Compostela, A Coruna
  - Novartis Investigative Site, Huelva, Andalusia
  - Novartis Investigative Site, Majadahonda, Madrid
  - Novartis Investigative Site, Las Palmas GC
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Valencia
- Novartis Investigative Site, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=3007

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All eligible participants were randomized via a validated Interactive Response Technology (IRT) to one of the treatment arms. Randomization was stratified by 2 factors: region, and ACEI/ARB or sacubitril/valsartan background treatment, respectively. Stratified randomization ensured that arms 1-4 had 1:2 ratio of participants on ACEI/ARB or sacubitril/valsartan background treatment, respectively, and arm 5 had only participants on prior ACEI/ARB background treatment.
Groups:
- XXB750 Placebo (Arm 1): XXB750 Placebo SC injection every 4 weeks during the randomized treatment period (Day 1, Week 4, Week 8 and Week 12)
- XXB750 60 mg (Arm 2): XXB750 60 mg SC injection every 4 weeks during the randomized treatment period (Day 1, Week 4, Week 8 and Week 12)
- XXB750 120 mg (Arm 3): XXB750 60 mg SC injection on Day 1 followed by XXB750 120 mg SC injection every 4 weeks during the randomized treatment period (Week 4, Week 8 and Week 12)
- XXB750 240 mg (Arm 4): No participants were exposed to the planned highest target dose of 240 mg
- Sacubitril/Valsartan (Arm 5): Participants switched from their pre-study ACEI/ARB treatment to open label tablet Sacubitril/valsartan, target dose 97/103 mg bid (Sac/Val)
Period: Overall Study
Arm/Group | XXB750 Placebo (Arm 1) | XXB750 60 mg (Arm 2) | XXB750 120 mg (Arm 3) | XXB750 240 mg (Arm 4) | Sacubitril/Valsartan (Arm 5)
Started | 29 | 26 | 56 | 0 | 25
Full analysis set (FAS) (All participants to whom study treatment has been assigned by randomization and who were not mis-randomized. Mis-randomized participants were those who had not been qualified for randomization, had been inadvertently randomized into the study and did not receive any study medication. According to the intent to treat principle, participants were analyzed according to the treatment they had been assigned to during the randomization procedure.) | 29 | 26 | 55 | 0 | 25
Safety set (SAF) (All randomized participants who received at least 1 dose of study treatment. Participants were analyzed according to the study treatment received, where treatment received is defined as the randomized/assigned treatment if the participant took at least 1 dose/injection of that treatment or the first treatment received if the randomized/assigned treatment was never received.) | 29 | 26 | 54 | 0 | 25
Completed | 9 | 6 | 16 | 0 | 3
Not Completed | 20 | 20 | 40 | 0 | 22
Not completed — Mis-randomized | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0
Not completed — Death | 0 | 1 | 3 | 0 | 1
Not completed — Study Terminated by Sponsor | 20 | 17 | 33 | 0 | 21
Not completed — Subject Decision | 0 | 1 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: To help guard the safety of study participants, randomization initially excluded the planned highest target dose of 240 mg XXB750 (i.e., arm 4). The study was terminated prematurely prior to the pre-planned early safety analysis due to an imbalance in worsening heart failure events among participants randomized to XXB750 60 mg and 120 mg. Thus, no participants were exposed to the planned highest target dose of 240 mg every 4 weeks.
Groups:
- Total: Total of all reporting groups
Arm/Group | XXB750 Placebo (Arm 1) | XXB750 60 mg (Arm 2) | XXB750 120 mg (Arm 3) | XXB750 240 mg (Arm 4) | Sacubitril/Valsartan (Arm 5) | Total
Number analyzed (Participants) | 29 | 26 | 55 | 0 | 25 | 135
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 16 | 0 | 12 | 43
  >=65 years | 22 | 18 | 39 | 0 | 13 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.7 (11.0) | 69.6 (9.7) | 70.1 (10.0) |  | 67.3 (11.6) | 69.8 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 14 | 0 | 10 | 41
  Male | 21 | 17 | 41 | 0 | 15 | 94
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 25 | 24 | 43 | 0 | 22 | 114
  Black or African American | 2 | 1 | 6 | 0 | 1 | 10
  Asian | 2 | 1 | 6 | 0 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Ratio to Baseline in NT-proBNP at Week 16
Description: Summary statistics for observed NT-proBNP values are reported: Geometric mean ratio to baseline at week 16 is calculated by the geometric mean of the ratio of the week 16 value to the baseline value. Baseline is defined as the value at randomization visit.
Time Frame: Baseline and week 16
Population: Full analysis set, which includes all participants to whom study treatment has been assigned by randomization, except for those who have not been qualified for this (and have therefore not received any study drug) but have been inadvertently randomized into the trial. Only participants with a value at both baseline and week 16 visit are included for calculating geometric mean change from baseline at week 16.
Measure: Geometric Mean (95% Confidence Interval); unit: unitless
Arm/Group | XXB750 Placebo (Arm 1) | XXB750 60 mg (Arm 2) | XXB750 120 mg (Arm 3) | XXB750 240 mg (Arm 4) | Sacubitril/Valsartan (Arm 5)
Number analyzed (Participants) | 28 | 21 | 45 | 0 | 21
unitless | 0.903 [0.696 to 1.172] | 1.021 [0.717 to 1.453] | 1.515 [1.147 to 2.001] |  | 0.701 [0.446 to 1.102]

2. Other Pre Specified Outcome: Baseline NT-proBNP Levels
Description: Baseline is defined as the NT-proBNP value at randomization visit.
Time Frame: Baseline
Population: Full analysis set. Only participants with a value at baseline visit are included
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | XXB750 Placebo (Arm 1) | XXB750 60 mg (Arm 2) | XXB750 120 mg (Arm 3) | XXB750 240 mg (Arm 4) | Sacubitril/Valsartan (Arm 5)
Number analyzed (Participants) | 29 | 26 | 54 | 0 | 25
pmol/L | 211.910 [142.532 to 315.058] | 163.501 [116.109 to 230.236] | 166.327 [132.519 to 208.761] |  | 186.753 [136.068 to 256.318]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 12 weeks post treatment, up to a maximum duration of 24 weeks.
Arm/Group | XXB750 Placebo (Arm 1) | XXB750 60 mg (Arm 2) | XXB750 120 mg (Arm 3) | Sacubitril/Valsartan (Arm 5)
All-Cause Mortality (participants affected / at risk) | 0/29 | 1/26 | 3/54 | 1/25
Serious Adverse Events (participants affected / at risk) | 1/29 | 8/26 | 18/54 | 3/25
Other Adverse Events (participants affected / at risk) | 13/29 | 16/26 | 24/54 | 12/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XXB750 Placebo (Arm 1) (N=29) | XXB750 60 mg (Arm 2) (N=26) | XXB750 120 mg (Arm 3) (N=54) | Sacubitril/Valsartan (Arm 5) (N=25)
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 5 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 2 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Death (General disorders and administration site conditions) | 0 | 0 | 0 | 1
Post cholecystectomy syndrome (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Endocarditis (Infections and infestations) | 0 | 0 | 1 | 0
Enterococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 1 | 0
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Movement disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 3 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | XXB750 Placebo (Arm 1) (N=29) | XXB750 60 mg (Arm 2) (N=26) | XXB750 120 mg (Arm 3) (N=54) | Sacubitril/Valsartan (Arm 5) (N=25)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 2 | 1
Cardiac failure (Cardiac disorders) | 0 | 4 | 7 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Salivary gland calculus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders and administration site conditions) | 1 | 1 | 1 | 0
Chest pain (General disorders and administration site conditions) | 0 | 1 | 1 | 0
Gait disturbance (General disorders and administration site conditions) | 0 | 1 | 0 | 0
Influenza like illness (General disorders and administration site conditions) | 0 | 1 | 0 | 0
Malaise (General disorders and administration site conditions) | 1 | 0 | 0 | 0
Pyrexia (General disorders and administration site conditions) | 0 | 1 | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 2 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 3 | 2 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 0 | 3
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 1 | 2 | 0 | 2
Breath sounds abnormal (Investigations) | 0 | 1 | 0 | 0
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 | 1 | 0 | 0
Protein urine present (Investigations) | 1 | 0 | 0 | 0
Folate deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Cerebral microangiopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 2 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 4 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2 | 1
Hypotension (Vascular disorders) | 2 | 4 | 7 | 6
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2024-02-23): https://cdn.clinicaltrials.gov/large-docs/83/NCT06142383/Prot_002.pdf
  • Statistical Analysis Plan (2024-12-04): https://cdn.clinicaltrials.gov/large-docs/83/NCT06142383/SAP_004.pdf